CLINICAL TRIAL: NCT04562051
Title: Stratified vs Routine Prophylaxis in Living Kidney Transplantation From HBsAg+ Donors to HBsAg- Recipients
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Director, West China Hospital
Other Study IDs: WestChina-KT
Record Dates: First submitted 2020-09-11; First posted 2020-09-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplantation; HBV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stratified prophylaxis group: The process of stratified prophylaxis was as follows. 1) If the recipient's HBsAb level is more than 100 IU/L and the donor is HBV DNA-, the recipient will not receive any preventive measures; 2) If the recipient's HBsAb is more than 100 IU/L and the donor is HBV DNA+, the recipient receives antiviral treatment for 1 month; 3) If the recipient's HBsAb is between 10 and 100 IU/L, the recipient is treated with single dose HBIG and antiviral treatment for 1 month regardless of the donor's HBV DNA status; 4) If the recipient's HBsAb is less than 10 IU/L, the recipient will receive single dose HBIG and antiviral treatment for 1 month regardless of the donor's HBV DNA status.
  Interventions: Other: prophylaxis regimen
- Routine prophylaxis group: Transplant centers adopted routine prophylaxis based on clinical experience
  Interventions: Other: prophylaxis regimen

INTERVENTIONS:
Other: prophylaxis regimen — All recipients were divided into two groups: stratified prophylaxis group based on donors' and recipients' characteristics and routine prophylaxis group based on clinical experience

SUMMARY:
This is a multicenter, prospective, observational study to compare the efficacy and safety of stratified prophylaxis based on donors' and recipients' risk factors vs routine prophylaxis bases on clinical experience in living kidney transplantation from HBsAg+ donors to HBsAg- recipients. The follow-up period was 2 years after renal transplantation. The primary outcome was prevention failure of HBV transmission (any one of HBsAg - → +, HBV DNA - → +, HBeAg - → +, HBeAb - → +, HBcAb - → +, active liver function damage and death in the recipient).

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with end-stage renal diseases and suitable for living kidney transplantation;
2. HBsAg+ donor was the only donor;
3. age and sex of donors and recipients were unrestricted;
4. ABO compatible or incompatible between the donor and recipient;
5. The living donor voluntarily donates one of their kidneys to the recipient free of charge;
6. The donor and recipient can understand the purpose and risk of living KT and sign informed consent;
7. Ethics committee approved.

Exclusion Criteria:

1. preoperative abnormal liver dysfunction in the donor or recipient (ALT > 60IU/L for females, and >75 IU/L for males; or total bilirubin > 34 umol/L); or preoperative ultrasonography in the donor or recipient reported hepatic cirrhosis;
2. positive complement-dependent cytotoxicity cross-match test;
3. combined HCV or HIV infection in the donor or recipient;
4. diagnosed with malignancy or had a history of malignancy in the past 5 years;
5. non-kidney transplantation history.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplantation from HBsAg+ donors to HBsAg- recipients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
composite outcome: prevention failure of HBV transmission from HBsAg+ donors to HBsAg- recipients | 2020.9-2025.10
  The primary outcome is the incidence of prevention failure of HBV transmission from HBsAg+ donors to HBsAg- recipients, which is a composite endpoint. The composite outcome includes HBsAg - → +, HBV DNA - → +, HBeAg - → +, HBeAb - → +, HBcAb - → +, active liver function damage and death in the recipients. Liver function damage is defined as postoperative abnormal liver dysfunction (ALT > 60IU/L for females, and >75 IU/L for males; or total bilirubin > 34 umol/L); or postoperative ultrasonography reported hepatic cirrhosis in the recipient.

SECONDARY OUTCOMES:
Graft loss | 2020.9-2025.10
  Graft loss was defined as re-establishment of long-term dialysis or estimated glomerular filtration rate (eGFR) of <15 ml/min.
biopsy-confirmed acute rejection | 2020.9-2025.10
  biopsy-confirmed acute rejection was diagnosed clinically based on a significant increase in serum creatinine levels of 50% or more within 3 days, which was not explained by other reasons and confirmed by biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Xianding Wang, MD, Study Director — Organ transplant center, Department of Urology, West China Hospital; Turun Song, MD, Principal Investigator — Organ Transplant Center, Department of Urology, West China Hospital; Yu Fan, MD, Principal Investigator — Organ Transplant Center, Department of Urology, West China Hospital; Zhongli Huang, MD, Principal Investigator — Organ Transplant Center, Department of Urology, West China Hospital; Saifu Yin, MB, Principal Investigator — Organ Transplant Center, Department of Urology, West China Hospital; Hongtao Liu, MD, Principal Investigator — The First Affiliated Hospital of USTC, University of Science and Technology of China; Wenjun Shang, MD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Honglan Zhou, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Tao Lin, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No